CLINICAL TRIAL: NCT05099731
Title: Evaluation of the Diagnostic Accuracy of aMMP-8 Point-of-care Test for the Discrimination of Periodontal Health and Disease Using Different Sampling Approaches: a Pilot Study Comparing Saliva and Oral Rinse
Brief Title: Diagnostic Accuracy of Matrix Metalloproteinase-8 Test for the Discrimination of Periodontal Health and Disease
Status: Completed | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Maurizio Tonetti, Professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: Pilotstudy0818
Record Dates: First submitted 2021-10-26; First posted 2021-10-29 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Periodontitis; Diagnostic Self Evaluation
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The application of point-of-care test with oral fluid-based biomarkers assisting in early-detection of gum disease is highly needed. Recently, a commercially available active Matrix metalloproteinase-8 (aMMP-8) point-of-care test (POCT) for detecting the risk of gum disease has been developed. Currently, there is a paucity of research to assess the performance of aMMP-8 POCT using different oral fluid sampling methods. This study will evaluate the accuracy of aMMP-8 POCT for discriminating periodontal health from disease in saliva and oral rinse.The information obtained from this study may help us understand better which sample is superior for the early detection of gum disease.

DETAILED DESCRIPTION:
The detection of the risk for periodontitis, one of the major global burdens of disease, prior to noticeable signs and symptoms is of great importance especially in non-dental settings. Oral fluids, including gingival crevicular fluid (GCF), saliva and oral rinse, have received considerable critical attention in the field of periodontal diagnostics for their non-invasive features and rich sources of biomarkers associated with the biological process in periodontal tissues. Saliva and oral rinse are preferred for screening purposes in a chair-side test, while GCF provides more site-specific information and has higher technical requirements.

Matrix metalloproteinases (MMPs) are a family of key host proteinases that regulate cell-matrix composition and MMP-8 is the main type of collagenases of MMP family responsible for collagen degradation of the periodontal supporting tissues. A growing body of evidence have indicated that elevated MMP-8, especially active form of MMP-8 (aMMP-8), has been detected in oral fluids of periodontitis (Kc et al., 2020). Currently, a commercially available aMMP-8 point-of-care test (POCT) has been developed (U.S. Patent No. 10,488,415, 2019). A recent study has assessed the diagnostic utility of this aMMP-8 POCT using oral rinse samples and showed moderate accuracy for detecting periodontitis (Deng et al., 2021). So far, however, there is a paucity of research to assess the performance of aMMP-8 POCT using different oral fluid sampling methods.

The study aims: i)to compare the diagnostic accuracy of aMMP-8 POCT for the discrimination of periodontal health and disease(s) in oral rinse and saliva; ii) to compare the diagnostic accuracy of aMMP-8 POCT for the discrimination of periodontal health and disease(s) in oral rinse during the first sampling and re-sampling.

This study is a cross-sectional diagnostic study.The whole study procedures will comprise the collection of different oral fluid samples, the conduction of aMMP-8 POCT using these samples (index test), followed by a routine full-mouth periodontal examination (reference standard). The details of the sequential study events include: 1) collection of unstimulated whole saliva sample by spitting method; 2) the first-time sampling of oral rinse (pure oral rinse); 3) re-sampling of oral rinse; 4) conduction of aMMP-8 point-of-care test using saliva and oral rinse samples collected at different times; and 5) routing full-mouth periodontal examinations to establish clinical case diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above
* Ability and willingness to give written informed consent

Exclusion Criteria:

* Edentulous mouth
* Pregnant females
* Having received professional periodontal treatment (other than supragingival cleaning) within the previous 12 months
* Having received antibiotic medication within the previous 3 months
* Presence of xerostomia interfering with saliva sampling
* Inability or unwillingness of individual to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consenting untreated patients seeking care at the Periodontology clinic and Implant Dentistry clinic of Shanghai Ninth People's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The area under the receiver operating characteristic curve (AUROC) measure | 1day
  Comparing the area under the receiver operating characteristic curve (AUROC) of aMMP-8 in different samples to correctly identify periodontitis cases at the time of completion of clinical examination

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial Implantology, Shanghai, Shanghai Municipality, China